CLINICAL TRIAL: NCT03781362
Title: A Phase 1, First-in-Human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of CPI-100 Via Intravenous Infusion in Patients With Advanced Solid Tumors
Brief Title: Study of CPI-100 in Patients With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coordination Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-CL18-001
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Advanced Tumors
Keywords: Intravenous infusion
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPI-100 Monotherapy (Experimental): Dose Escalation Groups:
  CPI-100 will be administered via intravenous infusion once every 2 weeks (Q2W) for up to 5 dose levels and once every 3 weeks (Q3W Arm A) for up to 4 dose levels in a 3 + 3 dose escalation study
  Dose Expansion Group: Maximum tolerated dose or the recommended Phase 2 dose (RP2D) from dose escalation group
  Interventions: Drug: CPI-100
- CPI-100 Combination with Capecitabine (Experimental): CPI-100 will be administered via intravenous infusion once every 3 weeks in combination with oral capecitabine for up to 4 dose levels in a dose escalation study (Q3W Arm B)
  Interventions: Drug: CPI-100; Drug: Capecitabine

INTERVENTIONS:
Drug: CPI-100 — CPI-100 will be administered via intravenous infusion on Day 1 of a 14-Day cycle
Drug: Capecitabine — Capecitabine will be administered 1000 mg/m2 orally twice a day for 2 weeks followed by a 7-day rest period
  Arms: CPI-100 Combination with Capecitabine

SUMMARY:
This is a prospective, open-label, 2-arm, non-randomized study of CPI-100 in patients with advanced tumors. CPI-100 is administered via intravenous infusion in a 3 + 3 study design to identify the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
Primary Objectives:

• To determine the safety, tolerability and maximum tolerated dose (MTD) of CPI-100 as once every two weeks (Q2W) and once every three weeks (Q3W) regimens in patients with advanced tumors

Secondary Objectives:

* To evaluate the pharmacokinetics (PK) of CPI-100
* To evaluate clinical response and resolution of symptoms after CPI-100 treatment
* To characterize adverse events of CPI-100 monotherapy and CPI-100 in combination with capecitabine in patients with advanced cancers

Up to 5 dose levels of CPI-100 Q2W, 4 dose levels of Q3W regimen of CPI-100 monotherapy (Q3W Arm A) and 4 dose levels of Q3W regimen of CPI-100 in combination with capecitabine (Q3W Arm B) will be tested in a dose escalation study. MTD will be defined as the dose associated with a dose limiting toxicity (DLT) in less than or equal to 33% of patients at the dose level tested. Dose limiting toxicity (DLT) is defined as one of the following events occurring from the intravenous injection of CPI-100 within 28 days (Q2W) or 42 days (Q3W):

* Grade 4 or greater treatment related adverse events
* Any Grade 3 or greater treatment related non-hematologic, non-dermatologic toxicity (including nausea, vomiting or diarrhea lasting more than 72 hours)

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically confirmed diagnosis of advanced solid tumor
* Have advanced or metastatic disease refractory to standard curative or palliative therapy or contraindication to standard therapy
* Be reasonably recovered from preceding major surgery or no major surgery within 4 weeks prior to the start of Day 1 treatment
* Have a negative pregnancy test for females with child bearing age at screening and should not be breast feeding
* Be willing to abstain from sexual activity or practice physical barrier contraception from study entry to 6 months after the last day of treatment

Exclusion Criteria:

* Have peripheral neuropathy of Grade 3 or Grade 4 at screening
* Have peripheral sensory neuropathy of Grade 2 or greater at screening
* Have an interval from previous neurotoxic drugs less than 3 months unless reasonably recovered from all grades of neurotoxicity to grade 1 or lower as judged by the investigator
* Have known hypersensitivity to chemotherapeutic agents
* Have a history of thrombocytopenia with complications including hemorrhage or bleeding > Grade 2 that required medical intervention or any hemolytic condition or coagulation disorders that would make participation unsafe
* Have unresolved toxicity from previous treatment or previous investigational agents; excluding alopecia
* Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Days
  • To determine the maximum tolerated dose (MTD), which is defined as the dose level at which fewer than 33% of patients experience a dose limiting toxicity (DLT) using a 3+3 strategy as assessed by CTCAE5

SECONDARY OUTCOMES:
Clinical Benefit | through study completion, an average of 4 months
  • To assess clinical benefit by response rate and resolution of symptoms, which will be reported as response rate (%)
Adverse Effect | through study completion, an average of 4 months
  • To assess adverse effect as either treatment-related or non-treatment-related as defined by CTCAE
Maximum Plasma Concentration (Cmax) | 8 Days
  • To evaluate maximum plasma concentration (Cmax) of CPI-100 in patients tested
Area Under the Curve (AUC) | 8 Days
  • To evaluate area under the curve (AUC) of CPI-100 in patients tested

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - South Texas Accelerated Research Therapeutics, Grand Rapids, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to confidentiality agreements